CLINICAL TRIAL: NCT01535404
Title: Right Versus Left Apical Transvenous Pacing for Patients With Preserved Left Ventricular Systolic Function (RIVELA) Study
Brief Title: Right Versus Left Apical Transvenous Pacing for Patients With Preserved Left Ventricular Systolic Function Study
Acronym: RIVELA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Haran Burri, MD (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor-Investigator, Haran Burri, MD, Assoc. Prof., University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRM-CH-Riv01
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2014-10

CONDITIONS: Bradyarrhythmia
MeSH Terms: conditions — Bradycardia | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right ventricular apex pacing (Active Comparator)
  Interventions: Device: Implantation procedure for a St-Jude Medical pacemaker system with right ventricular apex pacing
- Left ventricular apex pacing (Experimental)
  Interventions: Device: Implantation procedure for a St-Jude Medical pacemaker system with left ventricular apex pacing

INTERVENTIONS:
Device: Implantation procedure for a St-Jude Medical pacemaker system with right ventricular apex pacing — Implantation procedure for a St-Jude Medical pacemaker system with a transvenous ventricular and if applicable a right atrial lead
  Arms: Right ventricular apex pacing
Device: Implantation procedure for a St-Jude Medical pacemaker system with left ventricular apex pacing — Implantation procedure for a St-Jude Medical pacemaker system with a transvenous left ventricular (coronary sinus) and if applicable a right atrial lead
  Arms: Left ventricular apex pacing

SUMMARY:
The purpose of this study is to compare chronic (1-year) effects on left ventricular ejection fraction resulting from transvenous pacing of the right ventricular apex (RVA) versus the left ventricular apex (LVA) in patients with preserved or mildly reduced left ventricular systolic function (>= 45%).

DETAILED DESCRIPTION:
It is well established that chronic right ventricular apical pacing has an adverse effect on left ventricular systolic function. An alternative is pacing the left ventricular apex, which has shown more favourable results in terms of left ventricular pump function than the RVA in small series. The left ventricular apex may be paced via the coronary sinus tributary (e.g. in the anterior cardiac vein). Our study will compare effects of these two pacing sites on left ventricular ejection fraction measured by 3D-echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Requirement for ventricular pacing according to current guidelines (including chronic atrial fibrillation)
* Anticipated >=50% daily ventricular pacing
* LVEF >=45% as evaluated by 2D-echocardiography, 3D-echocardiography, magnetic resonance imaging or by radionuclide/contrast ventriculography
* Minimum age of 18 years, and at least 1 year life expectancy

Exclusion Criteria:

* Prior tricuspid valve replacement (annuloplasty is permitted)
* Intrinsic rhythm < 30bpm
* Patients with permanent atrial fibrillation who undergo ablation of the atrioventricular node.
* Echocardiographic window of insufficient quality for measuring LVEF
* Life expectancy of < 1year
* Pregnancy (women of childbearing potential will undergo pregnancy testing)
* Unable of unwilling to sign a patient informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduction in LVEF | baseline to one year

SECONDARY OUTCOMES:
Change in left ventricular end-systolic and end-diastolic volumes | one year
Dyssynchrony evaluation during RV and LV pacing | one year
Change in tricuspid regurgitation severity, if any | one year
Change in mitral regurgitation severity, if any | one year
Incidence of device-related complications | one year
Success rate of autocapture algorithm for left-and right-ventricular pacing | one year
Mortality and all cause hospitalization | one year
Reduction of LVEF at 1 year compared to baseline according to the following pre-specified subgroups: a) initial LVEF, b) gender, c)etiology (coronary artery disease, nonischemic cardiomyopathy) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Haran Burri, Assoc. Prof., Principal Investigator — University Hospital, Geneva; Angelo Auricchio, Prof., Principal Investigator — Fondazione Cardiocentro Ticino (Lugano); Christian Sticherling, Prof., Study Chair — University Hospital of Basel; Paul Erne, Prof., Study Chair — Luzerner Kantonsspital; Peter Ammann, PD Dr., Study Chair — Cantonal Hospital of St. Gallen; Frits Prinzen, Dr., Study Chair — Cardiovascular Research Institute, University of Maastricht
Locations (6):
- Cardiovascular Research Institute, University of Maastricht, Maastricht, Netherlands
- Switzerland (5):
  - University Hospital of Basel, Basel, Canton of Basel-City
  - University Hospital Geneva, Geneva, Canton of Geneva
  - Kantonsspital Luzern, Lucerne, Canton of Lucerne
  - Kantonsspital St-Gallen, Sankt Gallen, Canton of St. Gallen
  - Cardiocentro Ticino (Lugano), Lugano, Canton Ticino